CLINICAL TRIAL: NCT06263075
Title: Evaluation of the Hemodynamic Variability During Craniosynostosis Surgery: a Comparison Between Traditional Hemodynamic Monitoring and Pressure Recording Analytic Method (CRASY-PRAM)
Brief Title: Hemodynamic Monitoring During Craniosynostosis Surgery: Comparing Traditional and Newer Technology Monitors (CRASY-PRAM)
Acronym: CRASY-PRAM
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Maria Cristina Mondardini, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 717/2023/Oss/AOUBo; 6822 (Other: SirER (Emilia-Romagna Research Information System) platform)
Record Dates: First submitted 2024-01-22; First posted 2024-02-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Craniosynostoses; Hypovolemia; Hemorrhage; Hemodynamic Instability
Keywords: Monitoring Physiologic; Monitoring Intraoperative
MeSH Terms: conditions — Craniosynostoses; Hypovolemia; Hemorrhage | interventions — Monitoring, Intraoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants undergoing craniosynostosis corrective surgery: Infants aged 3 to 8 months with craniosynostosis admitted to the operating room of Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Azienda Ospedaliero-Universitaria (AOU) of Bologna Polyclinic Sant'Orsola to undergo corrective surgery.
  Interventions: Procedure: Intraoperative monitoring

INTERVENTIONS:
Procedure: Intraoperative monitoring — ANESTHESIOLOGICAL MANAGEMENT accords to usual practice. Participants underwent preoperative fasting (3 h for breast milk, 4 h for formula milk, and 1 h for clear liquids), no premedication, induction and maintenance by sevoflurane, fentanyl boluses for analgesia, mechanical ventilation (PEEP 4 cm H2O, target tidal volume 6-8 ml/Kg, end tidal CO2 32-40 mmHg), 10 ml/Kg/h of intraoperative fluids. Scalp block is performed before surgery.
  MONITORING DURING SURGERY: monitor devices routinely used are connected to the participant: Dräger Infinity Delta XL®, Masimo® for pulse oximetry (Rainbow SET), regional cerebral oximetry (O3TM), and (optional) brain function monitoring (Masimo® SedLine). Arterial blood gas test is sampled at the anesthesiologist's discretion. After the artery catheterization, the MostCare® system is simultaneously connected to the patient monitoring devices. Data are collected every 3 minutes, 6 minutes for the noninvasive blood pressure measurement.

SUMMARY:
Hemodynamic evaluation during pediatric anesthesia is essential to care management. Intraoperative cardiovascular instability is frequent in major surgeries, and appropriate monitoring is necessary to ensure safe anesthetic conduction and promptly detect changes in blood pressure, cardiac output, blood volume, and organ perfusion. In this context, advanced hemodynamic monitoring, continuous measuring, and estimating various parameters can allow a more specific hemodynamic profile and help identify the causal mechanisms of its variability. Moreover, the reference ranges of hemodynamic values in different pediatric ages and how to best monitor hemodynamic status in pediatrics are still debated.

Surgical treatment of craniosynostosis is usually performed at an early age, between 3 and 8 months of age. The operation is burdened by a high risk of hemodynamic instability related mainly, but not only, to potential substantial hemorrhagic losses.

This study aims to characterize the hemodynamic events occurring during corrective craniosynostosis surgery, recorded simultaneously with standard monitoring and Pressure Recording Analytic Method (PRAM), and to analyze the paired measurements.

DETAILED DESCRIPTION:
During major surgery under general anesthesia, the risk of hemodynamic instability and organ hypoperfusion resulting from depth of anesthesia, bleeding, or neurovegetative stimulation is high. In the pediatric age, it is essential to ensure adequate cerebral perfusion to preserve neurological function. Even more in younger age groups, given the limited knowledge of the safe boundaries of blood pressure and cerebral autoregulation, sufficient to ensure adequate cerebral perfusion. Traditional instrumental monitoring is clinically helpful but limited in specificity and accuracy. Instead, advanced hemodynamic monitoring techniques can allow early detection of changes in volemia and cardiac inotropism. The Pressure Recording Analytical Method (PRAM), installed in the monitor MostCare® (VYGON), analyzes the area under the curve of arterial blood pressure, beat by beat, to evaluate the dynamic impedance of the cardiovascular system. It estimates several parameters, including stroke volume and cardiac output, the preload by stroke volume variation and pulse pressure variation, the afterload by the systemic vascular resistances, and the arterial telesystolic elastance. Previous studies conducted on the pediatric population have demonstrated the applicability and reliability of MostCare® on young patients.

Craniosynostosis is an abnormal early fusion of cranial sutures. Physiological growth of the brain and impeded adaptation of the cranium will result in progressively increased intracranial pressure, dysmorphisms, delays, and impairment in neurodevelopment. Surgery is the core option for treatment, and the prognosis improves when performed soon, at 3-4 months of age or in the immediately following months. Hemodynamic changes resulting from deep anesthesia, bleeding, venous gas embolism, obstruction to cerebral venous outflow from an extreme head-bending position, and cerebrospinal fluid leakage after rupture of the dura may occur during the operation.

The objectives of the study are to describe and analyze the dynamic cardiovascular variables concurrently measured by MostCare® and other standardized monitors to capture events occurring in infants during corrective craniosynostosis surgery.

ELIGIBILITY:
Inclusion Criteria:

* Infants with craniosynostosis undergoing corrective surgery
* Ages between 3 and 8 months
* Physical status classification of the American Society of Anesthesiologists (ASA) </= 2
* Consent obtained from the patients' parents/legal guardians

Exclusion Criteria:

* Congenital or acquired cardiac disease
* Preoperative cardiac dysfunction
* Metabolic diseases
* Gestational age at birth <30 weeks
* Body weight less than 3 kg
* Dislocation or malfunction of the arterial catheter
* Malfunctioning of monitoring devices

Ages: 3 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Consecutive infants aged 3 to 8 months with craniosynostosis admitted to the operating room of IRCCS AOU of Bologna Polyclinic Sant'Orsola to undergo corrective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic events occurring during surgery | Entire duration of surgery
  Number of hemodynamic events during surgery. Hemodynamic events are defined as a reduction or increase of 20% from the baseline of parameters measured by monitors. The baseline value per individual participant corresponds to the value recorded for each parameter at the time of starting monitoring.

SECONDARY OUTCOMES:
Evaluation of changes in volemic status | during the surgery
  Absolute values and variations of Pulse Pressure Variation (PPV) from MostCare® every reduction of 20% from the baseline of invasive blood pressure (IBP).
Evaluation of changes in volemic status | during the surgery
  Absolute values and variations of Stroke Volume Variation (SVV) from MostCare® every reduction of 20% from the baseline of invasive blood pressure (IBP).
Evaluation of changes in systemic vascular resistance | during the surgery
  Absolute values and variations of Systemic Vascular Resistance Index (SVRI) from MostCare® every reduction of 20% from the baseline of invasive blood pressure (IBP).
Evaluation of changes in cardiac function | during the surgery
  Absolute values and variations of Cardiac output Index (CI) from MostCare® every reduction of 20% from the baseline of invasive blood pressure (IBP).
Evaluation of changes in cardiac function | during the surgery
  Absolute values and variations of maximum pressure variation (dP/dt (max) from MostCare® every reduction of 20% from the baseline of invasive blood pressure (IBP).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Mondardini, MD, Principal Investigator — IRCCS AOU of Bologna Policlinico Sant'Orsola
Locations (1):
- IRCCS AOU of Bologna Policlinico Sant'Orsola, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh Y, Villaescusa JU, da Cruz EM, Tibby SM, Bottari G, Saxena R, Guillen M, Herce JL, Di Nardo M, Cecchetti C, Brierley J, de Boode W, Lemson J. Recommendations for hemodynamic monitoring for critically ill children-expert consensus statement issued by the cardiovascular dynamics section of the European Society of Paediatric and Neonatal Intensive Care (ESPNIC). Crit Care. 2020 Oct 22;24(1):620. doi: 10.1186/s13054-020-03326-2. PMID 33092621
- [Result] Calabrese S, Angileri S, Paolicchi O, Mancinelli P, Colosimo D, Ricci Z. Noninvasive vs. invasive arterial pressure during pediatric non cardiac surgery. Minerva Anestesiol. 2023 Sep;89(9):841-842. doi: 10.23736/S0375-9393.23.17338-X. Epub 2023 May 9. No abstract available. PMID 37158631
- [Result] de Graaff JC, Pasma W, van Buuren S, Duijghuisen JJ, Nafiu OO, Kheterpal S, van Klei WA. Reference Values for Noninvasive Blood Pressure in Children during Anesthesia: A Multicentered Retrospective Observational Cohort Study. Anesthesiology. 2016 Nov;125(5):904-913. doi: 10.1097/ALN.0000000000001310. PMID 27606930
- [Result] Garisto C, Favia I, Ricci Z, Romagnoli S, Haiberger R, Polito A, Cogo P. Pressure recording analytical method and bioreactance for stroke volume index monitoring during pediatric cardiac surgery. Paediatr Anaesth. 2015 Feb;25(2):143-9. doi: 10.1111/pan.12360. Epub 2014 Feb 3. PMID 24491036
- [Result] Ricci Z, Pilati M, Favia I, Garisto C, Rossi E, Romagnoli S. Hemodynamic monitoring by pulse contour analysis in critically ill children with congenital heart disease. Pediatr Crit Care Med. 2011 Sep;12(5):608-9; author reply 609-10. doi: 10.1097/PCC.0b013e318219182b. No abstract available. PMID 21897172
- [Result] Meier N. Anesthetic Considerations for Pediatric Craniofacial Surgery. Anesthesiol Clin. 2021 Mar;39(1):53-70. doi: 10.1016/j.anclin.2020.10.002. Epub 2021 Jan 12. PMID 33563386